CLINICAL TRIAL: NCT05502159
Title: Comparison of Ultrasound-Guided M-TAPA Block and External Oblique Intercostal Block for Postoperative Analgesia Management in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: M-Tapa Block vs External Oblique Intercostal Block for Laparoscopic Cholesistectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 30
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cholecystitis; Cholecystitis, Acute
Keywords: Laparoscopic Cholesistectomy; Postoperative pain management; M-TAPA block; External oblique intercostal block
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic cholesistectomy surgery will be included in the study. Patients will be randomly divided into two groups (Group M = M-TAPA group, Group EOB = EOB group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA = M-TAPA group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 0,5 mg/kg meperidin will be performed for rescue analgesia.
  Interventions: Drug: M-TAPA
- Group EOB = EOB group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 0,5 mg/kg meperidin will be performed for rescue analgesia.
  Interventions: Drug: EOB

INTERVENTIONS:
Drug: M-TAPA — Under aseptic conditions, a high-frequency linear probe will be placed on the costochondral angle in the sagittal plane. Then the probe will be slightly angled deeply to visualize the lower view of the perichondrium. We will perform M-TAPA with total of 40 ml (20 ml for each side) of %0,25 bupivacaine.
  Arms: Group M-TAPA = M-TAPA group
Drug: EOB — In the supine position, a high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed on the midaxillary line between the spina iliaca anterior superior and the umbilicus. Using the In-Plane technique, 5 ml of saline will be injected under the external oblique muscle of the block needle and the block location will be confirmed. After the block location is confirmed, 20 ml of 0.25% bupivacaine will be administered. The same procedure will be applied to the other side (40 ml of 0.25% bupivacaine in total).
  Arms: Group EOB = EOB group

SUMMARY:
Ultrasound (US)-guided Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block is a novel block that provides effective analgesia in the anterior and lateral abdominal walls after laparoscopic surgery, and local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral wall and may be an opioid-sparing strategy with good quality recovery in patients undergoing laparoscopic surgery.

US-guided External oblique intercostal block (EOB) is a block performed by injection of local anesthetic between the external and internal oblique muscles. This block provides abdominal analgesia between T6-T10 levels. There are studies in the literature showing that it provides effective analgesia. However, there is no study comparing M-TAPA and EOB yet.

In this study, our aim is to compare the effectiveness of US-guided M-TAPA block and EOB for postoperative analgesia management after laparoscopic cholecystectomy surgery. Our primary aim is to compare patient recovery scores (QoR15 Turkish version), our secondary aim is to compare postoperative pain scores (24-hour NRS), postoperative rescue analgesic use (opioid), and opioid-related side effects (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Cholecystectomy is the most common of the abdominal surgical procedures performed in developed countries and is usually performed laparoscopically. Many factors play a role in the pain that develops after laparoscopic cholecystectomy and is generally considered to be visceral pain. Phrenic nerve irritation as a result of CO2 insufflation into the peritoneal cavity, abdominal distention, tissue trauma, trauma due to the removal of the gallbladder, sociocultural status, and individual factors are the factors that play a role in the emergence of this pain.

Postoperative pain is acute pain that is accompanied by an inflammatory process due to surgical trauma and gradually decreases with tissue healing. Postoperative pain in patients undergoing laparoscopic cholecystectomy is a serious problem that reduces patient comfort and delays the patient's return to work after surgery. Successful postoperative analgesia, occurs in the patient due to pain; It is a known fact that it prevents many of the effects such as not being able to breathe easily and delayed mobilization.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a new block that provides effective analgesia in the anterior and lateral abdominal walls after laparoscopic surgery in which local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral wall and may be an opioid-sparing strategy with good quality recovery in patients undergoing laparoscopic surgery.

M-TAPA block provides analgesia in the T5-T11 abdominal region. Sonoanatomy is easy to visualize on US and the spread of local anesthetic can be easily seen. With the cephalo-caudal spread of the local anesthetic solution, analgesia occurs in several dermatomes. In the literature, there are studies investigating the effectiveness of M-TAPA block for post-operative pain management in bariatric surgery. In the literature, there is no randomized study evaluating the effectiveness of M-TAPA block for postoperative analgesia management after laparoscopic cholecystectomy operation.

US-guided External oblique intercostal block (EOB) is a block performed by injection of local anesthetic between the external and internal oblique muscles. This block provides abdominal analgesia between T6-T10 levels. There are studies in the literature showing that it provides effective analgesia. However, there is no study comparing M-TAPA and EOB yet.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic inguinal hernia repair surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* anticoagulant treatment
* local anesthetics and opioid allergy
* Infection at the site of block
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | Change from baseline score at postoperative 24 hour
  We will use the Turkish version of Quality of Recovery / QoR-15 questionairre

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Postoperative 24 hours period (0, 2, 4, 8, 16 ve 24 h)
  Change from Baseline Pain Scores at Postoperative 24 hours.
The use of rescue analgesia | Postoperative 24 hours period
  Meperidin using (Number of Participants and Concentration of Meperidin)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Altiparmak B, Toker MK, Uysal AI, Turan M, Demirbilek SG. Reply to Tulgar et al.: Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:150-151. doi: 10.1016/j.jclinane.2018.12.005. Epub 2018 Dec 12. No abstract available. PMID 30553219
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Background] Hamilton DL, Manickam BP, Wilson MAJ, Abdel Meguid E. External oblique fascial plane block. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100256. doi: 10.1136/rapm-2018-100256. Online ahead of print. No abstract available. PMID 30635518
- [Background] Tulgar S, Ahiskalioglu A, Selvi O, Thomas DT, Ozer Z. Similarities between external oblique fascial plane block and blockage of thoracoabdominal nerves through perichondral approach (TAPA). J Clin Anesth. 2019 Nov;57:91-92. doi: 10.1016/j.jclinane.2019.03.027. Epub 2019 Mar 29. No abstract available. PMID 30933854